CLINICAL TRIAL: NCT00393809
Title: Phase 1/2a, Dose-Escalation, Safety and Proof of Concept Study of Intravesical DTA-H19 in Patients With Superficial Bladder Cancer
Brief Title: Safety and Proof of Concept Study of Intravesical DTA-H19 in Patients With Superficial Bladder Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hebrew University of Jerusalem (Other)
Collaborators: Anchiano Therapeutics Israel Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-05-02.CTIL
Record Dates: First submitted 2006-10-26; First posted 2006-10-30 (Estimated); Last update posted 2008-01-07 (Estimated); Status verified 2007-12

CONDITIONS: Bladder Neoplasms
Keywords: transitional cell carcinoma; H19 gene; plasmid; diphtheria toxin
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell

INTERVENTIONS:
Drug: DTA-H19

SUMMARY:
This study is designed to assess the safety and preliminary efficacy of five different doses of DTA-H19 given as six intravesical infusions into the bladder of patients with superficial bladder cancer who have failed intravesical therapy with Bacille Calmette-Guérin (BCG).DTA-H19 is a DNA plasmid that contains H19 gene regulatory sequences that drive the expression of an intracellular toxin [diphtheria toxin A (DTA) chain]only in cancer cells and not in normal cells. In line with the standard procedure for DNA plasmid pharmaceutical products, another chemical component will be added to the solution, called PEI (polyethlenimine) in a liquid solution, which improves the ability of the DNA plasmid to enter the cells.

DETAILED DESCRIPTION:
This study is designed to assess the safety and preliminary efficacy of five different doses of DTA-H19 given as six intravesical infusions into the bladder of patients with superficial bladder cancer [stages Ta and carcinoma in situ (CIS)] who have failed intravesical therapy with Bacille Calmette-Guérin (BCG). The primary safety outcome measure is the maximum tolerated dose (MTD). DTA-H19 is a DNA plasmid that contains H19 gene regulatory sequences that drive the expression of an intracellular toxin [diphtheria toxin A (DTA) chain]. This is a Patient-Oriented, Targeted Therapy as DTA expression is triggered by the presence of H19 transcription factors found only in bladder tumor and not normal bladder cells.

A maximum of 18 patients with histologically confirmed H19 positive superficial bladder cancer with multiple or recurrent stage Ta tumors or CIS will be included in this study. Patients with any grade 3, or any stage T1 or higher stage, will be excluded. This is a multicenter, dose escalation study in which, after eligibility criteria have been met, patients in five groups of 3 patients each, will receive escalating doses of DTA-H19 intravesically over a seven-week period. Treatments will be given weekly for three weeks followed one week later by safety and disease assessments, then another 3 weekly instillations will be performed. Each dose cohort will receive the same dose for all treatments. The first dose cohort will receive 2 mg of DTA-H19 plasmid per intravesical treatment for all treatments. The next dose cohort of 3 patients will receive 4 mg, the next 6 mg, the next 12 mg,and then the final dose cohort will receive 20 mg of DTA-H19 plasmid DNA. All doses will be mixed with polyethylenimine (PEI) to improve transduction efficiency. Doses will be escalated if none of the first three patients in the preceding dose cohort experience a dose limiting toxicity (DLT) after the first three weekly intravesical treatments.

Clinical responses will be assessed 4, 8, and 12 weeks after the start of treatment. If the stage Ta marker lesion is still present at the week 12 assessment, it will be resected by transurethral resection (TUR). Patients whose disease has not progressed (i.e., no new lesions, increase in the size of the marker lesion, by at least 50%, or increase in stage or any grade 3) will be offered continued once monthly treatments and follow-up for up to one year

ELIGIBILITY:
Inclusion Criteria:

* Patients must have superficial transitional cell carcinoma of the bladder (stages Ta and/or CIS)
* Tumor biopsies must be shown to be positive for H19 gene by in situ hybridization
* Patients must have failed intravesical treatment with BCG

Exclusion Criteria:

* Patients with grade 3, or Stage 1 or higher stage TCC of the bladder
* Patients with any other malignancy that might impact 5-year survival or might be potentially confused with TCC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-01; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD)

SECONDARY OUTCOMES:
The percentage increase or reduction in the area of marker lesions
The number of patients with progressive disease
The time to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Sidi, MD, Principal Investigator — E. Wolfson Medical Center; Ilan Leibovitch, MD, Principal Investigator — Meir Medical Center
Locations (2):
- Israel (2):
  - E. Wolfson Medical Center, Holon
  - Meir Medical Center, Kfar Saba